CLINICAL TRIAL: NCT07026617
Title: Effectiveness of Adding Low Level Laser Therapy to Rocabado's Approach for Myogenic Temporomandibular Joint Disorders: A Double-Blind Placebo-Controlled Clinical Trial
Brief Title: Low Level Laser Therapy and Rocabado's Approach for Myogenic TMJ Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Shafiek Mustafa Saleh, assistance professor doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LLLT and myogenic TMJ
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Myogenic Temporomandibular Joint Disorders
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: Rocabado's approach in addition to LLLT
- control group (Placebo Comparator)
  Interventions: Other: control group

INTERVENTIONS:
Other: Rocabado's approach in addition to LLLT — The patients will recieve Rocabado's non-thrust manipulation: Non-thrust temporo-mandibular joint manipulations consisted of medial glide, lateral glide and anterior glide as described by Rocabado. Each glide was given for 10-15 repetitions for 5-6 times in a session. The grade of mobilization was beginning with Grade-1 or 2 and progressed to Grade-4 depending on subject condition. Total duration of mobilization was lasted for 20 minutes. in addition to low power gallium aluminum arsenide (GaAlAs).
  Arms: study group
Other: control group — The patients will recieve Rocabado's non-thrust manipulation: Non-thrust temporo-mandibular joint manipulations consisted of medial glide, lateral glide and anterior glide as described by Rocabado. Each glide was given for 10-15 repetitions for 5-6 times in a session. The grade of mobilization was beginning with Grade-1 or 2 and progressed to Grade-4 depending on subject condition. Total duration of mobilization was lasted for 20 minutes. in addition to lplacebo ow power gallium aluminum arsenide (GaAlAs).
  Arms: control group

SUMMARY:
Rocabado's 6x6 exercises are designed to improve muscular co-ordination, relax tense muscles, increase temporomandibular joint (TMJ) ROM, alter the jaw closure pattern and muscle strength. These exercises have been found to be beneficial in reducing pain and increasing masticatory muscle function, as well as restoring restricted joint mobility, muscle length limitation, and postural and functional limitations. In addition, low level laser therapy (LLLT) has been reported to reduce inflammation and pain in patients with TMJ dysfunction. Although that to the best of the authors' knowledge the combined effect of Rocabado's approach with LLLT has not been studied. So, the current study is the first double-blind placebo-controlled clinical trial that investigating the effect of adding LLLT to Rocabado's approach for TMJ myogenic disorders.

ELIGIBILITY:
Inclusion Criteria:

(1) The patient's ages ranged from 18 to 40 years ; (2) having symptoms of TMD for at least twelve weeks duration established by expert physician or orthopaedician; (3) mouth opening < 25mm

Exclusion Criteria:

(1) TMJ fracture undergone any surgical procedure for TMJ; (2) Fracture surrounding TMJ; (3) Dislocation or subluxation of TMJ; (4) Systemic generalized joint diseases, such as rheumatoid arthritis, and osteoporosis, congenital diseases or facial paralysis; (5) recently any dental treatment taken or surgery over TMJ; (6) Hematological cervical disorders which may affect the jaw; (7) Neurological deficits e.g. Bells palsy, Trigeminal neuralgia; (8) Recent infections (within the last six months) affecting the head and neck e.g. bone infections, meningitis, encephalitis, malaria, ear infection; (9) Participants who were using any functional appliances e.g. dentures, braces, bite appliances which had been adjusted or fitted in the last 12 weeks prior to the commencement of this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain pressure threshold of masticatory muscles | change from base line at 6 weeks.
  The pain pressure threshold over the temporalis and masseter muscles will be assessed using an algometer with a 1 cm2 probe tip (FDIX Digital Force Gage; Wagner Instruments).

SECONDARY OUTCOMES:
Assessment of Temporomandibular joint ROM | change from base line at 6 weeks.
  A therabite will be used to measure mandibular opening
Assessment of the function of Temporomandibular Joints | change from base line at 6 weeks.
  Temporomandibular Disorder Disability Questionnaire will be used for evaluating the temporomandibular joint function. It consists of the following subsections: the Temporomandibular Disorder Disability Index, Temporomandibular Disorder symptom intensity scale, and Temporomandibular Disorder symptom frequency scale.
Assessment of pain intensity using Numerical Rating Scale | change from base line at 6 weeks.
  in the rating scale the patient will be asked to indicate a number between 0 and 100 on a horizontal line, that best described his/her perceived level of pain intensity when it is at its worst and when it is at is least.